CLINICAL TRIAL: NCT05274477
Title: Randomized Placebo-controlled Phase II Cross-over Study on the Influence of Fampridine on Working Memory in Individuals With Post COVID-19 Condition With Subjective Cognitive Impairment
Brief Title: Influence of Fampridine on Working Memory in Individuals With Post COVID-19 Condition With Subjective Cognitive Impairment
Acronym: FamC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment difficulties
Sponsor: Prof. Dominique de Quervain, MD (Other)
Collaborators: Clinical Trial Unit, University Hospital Basel, Switzerland (Other); University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor-Investigator, Prof. Dominique de Quervain, MD, Director Division of Cognitive Neuroscience,, University of Basel
Organization: University of Basel (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2022-00452
Record Dates: First submitted 2022-03-03; First posted 2022-03-10 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Working Memory; Post-covid-19
MeSH Terms: interventions — 4-Aminopyridine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fampridin SR (Experimental): Active study medication consists of 7 tablets of fampridine SR 10 mg formulated for oral administration taken in the morning and evening 12 h apart without food. Tablets must be administered whole.
  There will be a washout period of at least 8 days equaling over 30 half-lives of the active substance fampridine (t½ = 6 h) between experimental and control intervention and up to 26 days depending on the individual scheduling of each subject.
  Interventions: Drug: Fampridine SR
- Placebo (Placebo Comparator): Identically looking placebo tablets consisting of widely identical additives formulated for oral administration.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fampridine SR — Fampridine SR is an inhibitor of voltage gated potassium channels and is approved in Switzerland for treatment of gait problems in patients with Multiple Sclerosis (MS).
  Arms: Fampridin SR
Drug: Placebo — no active component
  Arms: Placebo

SUMMARY:
In genome-wide association studies we identified potassium channels to be genetically linked to performance and neural activity of working memory in healthy humans. Furthermore, there is evidence in rodents and non-human primates that pharmacological blockade of potassium channels can improve working memory.

In the present study, we aim at investigating the effects of 10 mg fampridine (4-Aminopyridine), a potassium channel-blocking agent, on working memory performance in individuals with Post-COVID-19-Condition with subjective cognitive impairment. The hypothesis is that fampridine improves working memory performance.

Fampridine, especially its slow-release formulation (Fampyra®) is generally a safe drug with well-studied pharmacokinetic properties. It crosses the blood-brain barrier and reaches maximum concentration in the brain approximately 3.5h after single-dose administration. Evidence suggests that fampridine improves walking speed in patients with multiple sclerosis (MS), which led to FDA and EMA approval for this indication. The mode of action by which fampridine improves walking speed is probably its blockade of a spectrum of potassium channels that are exposed in demyelinated axons, leading to mitigation of potassium leakage and normalization of nerve conduction. Additionally, an action of fampridine at central synapses and increase of neurotransmitter release has been discussed.

ELIGIBILITY:
Inclusion Criteria:

* male or female;
* a valid positive PCR test or a documented certified rapid antigen test or a virus-specific antibody (nucleocapsid) test for COVID-19 issued at least 3 months prior to study;
* Above medium subjective working memory impairment (at least "much worse" in item 1a part 2 (cognitive abilities) of the Covid-Q screening questionnaire;
* present at least 3 months after COVID-19 infection and lasting for at least 2 months. (The impairment must have emerged after COVID-19 infection and cannot be explained by an alternative diagnosis);
* normotensive (BP: 90/60mmHg - 140/90mmHg);
* BMI: 19.0 - 40.0 kg/m2;
* Age: 18 - 69 years;
* fluent German-speaking;
* IC as documented by signature.

Exclusion Criteria:

* initiation of pharmacological treatment or change of dose within the 30 days preceding the present study
* contraindications to the class of drugs under study, e.g. known hypersensitivity or allergy to 4-aminopyridine
* use of potassium channel blockers within the last 3 months
* concomitant treatment with OCT 2 inhibitors and -substrates (e.g. cimetidine, propranolol)
* acute or chronic psychiatric disorder (e.g. major depression, psychosis, somatoform disorder, suicidal tendency)
* acute cerebrovascular condition
* history of seizures
* risk of lowered seizure threshold (due to e.g. sleep deprivation, withdrawal of alcohol after alcohol abuse)
* renal impairment
* history of malignant cancers
* walking problems (e.g. due to dizziness)
* other clinically significant concomitant disease states that could pose a safety risk (e.g. hepatic dysfunction, cardiovascular disease, urinary tract infection)
* bradycardia < 50/min during clinical examination
* clinically significant laboratory or ECG abnormality that could be a safety issue in the study
* known or suspected non-compliance (e.g. missing more than one dose of study medication per intervention phase)
* drug or alcohol abuse
* inability to follow the procedures of the study, e.g. due to language or psychological problems of the participant
* participation in another study with an investigational drug within the 30 days preceding and during the present study
* enrolment of the investigator, his/her family members, employees and other dependent persons
* pregnancy or breast feeding
* Intensive care treatment due to COVID-19 infection.

Exclusion Criteria concerning TMS measurement

* metal in the brain, skull or elsewhere in the body (e.g., splinters, fragments, clips, etc.)
* implanted neurostimulator (e.g., DBS, epidural/subdural, VNS)
* cardiac pacemaker or intracardiac lines
* medication infusion device
* piercings in the head area, pivot teeth (retainers are no exclusion criterion)
* tattoos (in the head area) with metallic inks or newly stung tattoos (< 3 months), as newly stung tattoos can be damaged by a magnetic field;
* condition after neurosurgery
* hearing problems or tinnitus
* not able to sit still due to tremor, tics, itching
* History of repeated syncope
* head trauma diagnosed as concussion or associated with loss of consciousness
* diagnosis of epilepsy, or a convulsion or a seizure in the past of the participant or his family
* TMS in the past showing problems
* MRI in the past showing problems
* surgical procedures to spinal cord
* spinal or ventricular derivations TMS measurement is optional. If a participant is eligible for the study, but prefers not to undergo TMS measurement or meets one or more exclusion criteria for TMS measurement, the participant can nevertheless be included in the study without rMT measurement using TMS.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2022-06-28 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Digits Span backward performance | first and last day of 3.5-days-treatment periods (each 4 hours after intake in the morning); to assess changes between the verum and placebo condition
  The Digit Span task is a subtest of an intelligence test for adults ("Wechsler Intelligenztest für Erwachsene" (WIE; (von Aster 2006)). Total scores for digit span backward will be calculated as described in the manual of the WIE. Minimum 0 points and maximum 12 points. Parallel version will be used for the altogether four assessments at the beginning (visits 2 and 4) and at the end (visits 3 and 5) of both treatment phases.

SECONDARY OUTCOMES:
Digits Span forward performance | first and last day of 3.5-days-treatment periods (each 4 hours after intake in the morning); to assess changes between the verum and placebo condition
  The Digit Span task is a subtest of an intelligence test for adults ("Wechsler Intelligenztest für Erwachsene" (WIE; (von Aster 2006)). Total scores for digit span backward will be calculated as described in the manual of the WIE. Minimum 0 points and maximum 12 points. Parallel version will be used for the altogether four assessments at the beginning (visits 2 and 4) and at the end (visits 3 and 5) of both treatment phases.
Red Button Task | first and last day of 3.5-days-treatment periods (each 4 hours after intake in the morning); to assess changes between the verum and placebo condition
  Reaction time test (Red Button Task), adapted from (Dinges and Powell, 1985): participant sits in front of a screen showing a gray circle in the middle of the screen. The circle's color turn into red and participant will be instructed to push a button as soon as the color changes. The period between the time of color change and button push is measured in miliseconds and will be considered as reaction time.
Symbol Digit Modalities Test, SDMT | first and last day of 3.5-days-treatment periods (each 4 hours after intake in the morning); to assess changes between the verum and placebo condition
  Symbol Digit Modalities Test, SDMT (Smith 2013, 13th edition), a processing speed test. The test consists of the presentation of a series of 9 symbols, each of them is paired with a single digit, labelled 1-9, in a key at the top of a sheet. The remainder of the page has a pseudorandomized sequence of the symbols and the participant must respond with the digit associated with each of these as quickly as possible. The score is the number of correct answers in 90 seconds. The administration of SDMT will be preceded by a learning sequence at both timepoints. It will be used parallel versions for all test days.
Verbal episodic memory performance (word list) | first and last day of 3.5-days-treatment periods (each 4 hours after intake in the morning); to assess changes between the verum and placebo condition
  Verbal episodic memory performance (15 words) measured by immediate and delayed word-list recall. Adapted from a subtest of the German test called "Verbaler Lern- und Merkfähigkeits-Test" (VLMT; Helmstaedter/Lendt/Lux, 2001).
Lexical ability | first and last day of 3.5-days-treatment periods (each 4 hours after intake in the morning); to assess changes between the verum and placebo condition
  Lexical ability measured by phonemic fluency test after acute and repeated intake of study medication (S-words); adapted from a subtest of the German test called "Regensburger Wortflüssigkeits-Test" (RWT; Aschenbrenner/Tucha/Lange, 2001). In this task participants should name orally as many words as possible initiating with a special letter in one minute (e.g. Mary, Milk, Mouse, etc. for the letter M) the number of unique meaningful words will be considered as the participant's score.
Bochumer Matrizentest (BOMAT - standard) | first and last day of 3.5-days-treatment periods (each 4 hours after intake in the morning); to assess changes between the verum and placebo condition
  Fluid intelligence (Gf) will be measured with the Bochumer Matrizentest (BOMAT - standard; Hossiep/Hasella, 2010, 1st edition), matrix reasoning. BOMAT - standard consisting of 30 items will be administered. Parallel version will be used for the altogether four assessments at the beginning (visits 2 and 4) and at the end (visits 3 and 5) of both treatment phases. To create four versions, the original BOMAT versions A and B have been divided each into two versions (every second item) with 15 items each. A time-limited version (10 minutes) will be used to avoid a ceiling effect. The total score is calculated by summing the correct solutions, ranging between 0 to 15.
Subjective cognitive impairment | during the three 3 days of the treatment phase as compared to the 3 days before treatment; to assess changes between the verum and placebo condition
  Subjective cognitive symptoms are assessed with a self-administered questionnaire at the end of both treatment phases (visits 3 and 5). The participants are asked to rate the changes of cognitive abilities during the three 3 days of the treatment phase as compared to the 3 days before treatment on a 7 point likert scale (much worse - (…) - unchanged - (…) much better).This questionnaire contains questions about several domains of cognitive function (working memory, episodic memory, attention and concentration, executive function, lexical ability).
Resting motor threshold (rMT) | test days 2 and 4 (last day of treatment periods; approx. 5 hours after last intake of fampridine SR) to assess differences between the verum and placebo condition
  The resting motor threshold (rMT) will be measured by transcranial magnetic stimulation (TMS). rMT will be determined by measuring the motor evoked potential (MEP) in the abductor digiti

CONTACTS AND LOCATIONS:
Overall Officials: Dominique de Quervain, Prof. MD, Study Chair — University of Basel, Transfaculty Research Platform; Andreas Papassotiropoulos, Prof. MD, Study Chair — University of Basel, Transfaculty Research Platform
Locations (1):
- University of Basel, Transfaculty Research Platform, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
All IPD (de-identified) that underline results in a publication will be shared upon reasonable request.
Supporting Information: Study Protocol, SAP
Time Frame: IPD will be available after publication, study protocol (including statistical analysis plan) will be made available before start of the study.
Access Criteria: All IPD (de-identified) that underline results in a publication will be shared upon reasonable request for scientific purposes. A reasonable request consists of a short description of the scientific purpose. Request will be reviewed by the team of the principal investigator.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-04): https://cdn.clinicaltrials.gov/large-docs/77/NCT05274477/Prot_SAP_006.pdf